CLINICAL TRIAL: NCT01662622
Title: Minimal Alveolar Concentration of Sevoflurane Inducing Isoelectric Electroencephalogram
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Ministry of Health, China (Other Government); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Wei Mei, AssociateProfessor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJMZK20120301
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Middle Aged Patients; Sevoflurane; General Anesthesia
Keywords: anaesthesia; middle aged; minimal alveolar concentration; sevoflurane; isoelectric EEG
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sevoflurane (Experimental): Anaesthesia was induced by 8% sevoflurane. Cisatracurium 0.15mg kg-1 was administered after loss of the lash reﬂex, then ventilated manually until the amplitude of T1 decreased to 0. Intubation was performed and switched to mechanical ventilation with a fresh gas flow 2L min-1. Gas concentrations were analysed using a gas analyser.The end-tidal concentration of carbon dioxide was maintained at 4.7kPa; an esophageal temperature probe was inserted and a warming unit was used if necessary to maintain normothermia (35.5°-38.5°). The surgical incision was performed at least 30min after tracheal intubation. When arterial blood pressure (MAP) decrease exceeding 20% of baseline values. Phenylephrine 0.1mg was administered intravenously if necessary to maintained MAP and recorded.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — The design of experiment is referred to the "Dixon up-and-down" method. The first subject was designed to receive end-tidal sevoflurane concentration of 1.7%. For each subject, 30 min interval time was given. The isoelectric EEG was considered as significant when the isoelectric state last for more than 1min. The maximal burst suppression rate was recorded if isoelectric EEG was not reached. Heart rate and MAP, were recorded 2 and 1min before and 3 min after skin incision. Adrenergic reflexes positive cases were counted.

SUMMARY:
Sevoflurane can abolish movement or adrenergic response to noxious stimulus. In order to investigate the effect of sevoflurane on cerebral electrical activity, we determined the MAC of sevoflurane inducing isoelectric electroencephalogram (EEG) in 50% of the subjects (MACie) in middle aged subjects.

DETAILED DESCRIPTION:
Patients received sevoflurane for anesthesia induction and maintenance at preselected concentrations according to an 'up and down' design, with 0.2% as a stepsize. General anesthesia was induced and maintained with sevoflurane, tracheal intubation was facilitated with cisatracurium. After a steady-state period of 30min without surgical stimulation, the state of isoelectric EEG was considered as significant when a burst suppression ratio of 100% last for more than 1 min. The haemodynamic responses to skin incision and the vasopressor requirement to maintain cardiovascular system were also analysed according to the EEG state.

ELIGIBILITY:
Inclusion Criteria:

* 45-65yr
* upper abdominal surgery in general anaesthesia
* ASA physical status classification of I or II

Exclusion Criteria:

* neurological disease
* received central nervous system-active drugs
* cardiac ejection fraction less than 40%
* history of difficult intubation or anticipated difficult intubation
* daily alcohol consumption
* obesity, defined as a body-mass index of more than 30
* without informed consent

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
MACie | 30min
  Minimal Alveolar Concentration of sevoflurane inducing isoelectric electroencephalogram (EEG) in 50% of the subjects (MACie)

SECONDARY OUTCOMES:
MACbs | 30 min
  Minimal Alveolar Concentration of sevoflurane inducing inducing burst suppression EEG (MACbs) in middle aged adults.

OTHER OUTCOMES:
Hemodynamic parameters | 3 min
  Hemodynamic parameters 2 min before and 3 min after skin incision
Use of phenylephrine | 30 min
  Use of phenylephrine during induction and maintenance of anesthesia with sevoflurane.

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, MD., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China